CLINICAL TRIAL: NCT03404934
Title: A Multicenter Non-randomized Controlled Study (NRS) Evaluating the Use of Adaptive Anastomosis (CREX) in Clinical Practise
Brief Title: Clinical Study Verifying C-REX LapAid in Clinical Practice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by mutual agreement between the site and sponsor
Sponsor: Carponovum AB (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREX-005
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Cancer Colonic
Keywords: Adaptive anastomosis; C-REX; Colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-REX group (Experimental): After resection of the disease in colon, the intestinal ends will be anastomosed by the investigational device, i.e. C-REX LapAid and C-REX DMH/DMHC included in the C-REX Ring-locking Procedure.
  Interventions: Device: C-REX Ring-locking Procedure

INTERVENTIONS:
Device: C-REX Ring-locking Procedure — The C-REX Ring-locking Procedure is a method based on adaptive anastomosis, in which intestinal ends adapt to each other after resection due to tumor, injury, or other disease.
  The investigational devices comprised of two components, i.e. C-REX LapAid and C-REX DMH/DMHC

SUMMARY:
In colorectal surgery, hand suturing and stapling are routine methods for performing intestinal anastomoses, and these methods appear to be similar in terms of clinical safety. Despite several years of experience with surgical procedures as well as improvements to the medical devices, problems with disturbed anastomotic healing leading to leakage and stenosis after colorectal surgery remain a significant challenge for surgeons. A frequency of anastomotic leakage after stapling or suturing has been reported to range from 3% to 20%. In addition, preoperative radiotherapy has been shown to increase the risk of anastomotic leakage even further.

The methods that are used today to detect leakages are unfortunately inaccurately and limited to monitoring symptoms, temperature, CRP-levels, and performing abdominal examinations and CT-scans. These clinical signs and parameters usually become apparent several days after onset of the leakage, which leads to a delayed diagnosis. Anastomotic leakage is not only a significant cause of increased morbidity of complications and mortality in patients, but also associated with increased risk of local recurrence and poor prognosis. Moreover, when reoperation is required to fix the leakage, a permanent stoma may be made at the level of the sigmoid colon and this procedure impacts live quality of patients negatively.

Based on the above considerations, a novel, adaptive anastomotic method has been developed by CarpoNovum to achieve a safer anastomosis. The method's working name is C-REX Ring-locking Procedure. C-REX is referred to our Colorectal anastomotic rings for Re-join the intestinal ends and validate the anastomosis, with function of Extract samples for analysis and conduct X-ray through connected catheters.

The novel adaptive anastomotic medical devices, C-REX LapAid and C-REX DMH/DMHC are easy to use, with unique possibility to control the anastomosis during and after surgery. The previous successful preclinical study encourages a clinical verification in patients undergoing colonic resection to evaluate the safety and performance of C-REX Ring-locking Procedure by use of C-REX LapAid and C-REX DMH/DMHC.

DETAILED DESCRIPTION:
OVERALL DESIGN The study is a prospective, multicenter, single arm study Possible study candidates are patients requiring resection of the left colon (descending colon and sigmoid) or the upper rectum (15cm above the anal rim) due to malign or benign disease. After informed consent has been achieved, and after physical examination and checking of inclusion/exclusion criteria, potential subjects will be enrolled in the study, and the investigational surgery will be performed during hospitalization. The devices, i.e. C-REX LapAid and C-REX DMH/DMHC, included in C-REX Ring-locking Procedure are applied to the inside of the intestine and connected to catheters that allow monitoring of the anastomosis (if DMC is applied).

The healing period is expected to be approximately 10 ± 2 days. The short-term implant, i.e. the anastomotic ring, detaches via necrosis on the inner part of the intestinal surface and is expelled the natural way during hospitalization.

The subject can be discharged from the hospital when the short-term implant has been evacuated, and the subject has begun to eat and has normal bowel movements. The observation period lasts until 30 days after surgery. The subject then continues follow-up according to local routine.

QUALITY CONTROL Authorization to perform C-REX Ring-locking Procedure According to CarpoNovum's regulation (Document 0041: Procedure, Accreditation of Surgeons for Clinical Studies), clinical investigators must be authorized to conduct the C-REX Ring-locking Procedure with C-REX LapAid and C-REX DMH/DMHC by performing at least one surgery on pigs and at least one train-in surgery on patients with the person in charge of the study (MD, PhD, Senior colorectal surgeon Anders Grönberg). When the clinical investigator is authorized to perform the C-REX Ring-locking Procedure with C-REX LapAid System, he or she receives a certificate. This certificate could also admit the clinical investigator the right to authorize other surgeons to perform C-REX Ring-locking Procedure with C-REX LapAid and C-REX DMH/DMHC (i.e. to perform at least one operations on pigs and at least one train-in operations on patients with the authorized clinical investigator).

Monitoring To ensure that the study is appropriately conducted, a monitor appointed by the sponsor will visit the investigation site regularly and oversee the investigator's compliance with the CIP, perform source-data verification and report to the sponsor on the progress of the study.

Each investigation site and clinical investigator in the study will be monitored. On all occasions, the responsible monitor and/or the person in charge of the study will secure for example that:

1. Compliance with CIP is maintained and any deviation from CIP is discussed with the clinical investigators, documented and reported to the sponsor; if the changes are significant, the competent authority and the ethical committee will be informed;
2. The device is being used according to CIP, IB and IFU, and if modifications are required either to the device or its method of use or to the CIP, this need shall be reported to the sponsor;
3. Signed and dated informed consent forms have been obtained from each subject at the time of enrolment and before any study-related procedures are undertaken;
4. The data in CRFs are complete, are recorded in a timely manner and are consistent with the source data;
5. Traceability and device accountability of the investigational device are properly maintained;
6. Maintenance and calibration of equipment relevant for assessment of the study is performed;
7. Possible adverse events or device deficiencies have been properly documented and reported;
8. Subjects withdrawal and/or non-compliance is documented and discussed with the clinical investigator and reported to the sponsor;
9. Clinical investigators have and continue to have staff and facilities to conduct the study safely and effectively;
10. Clinical investigators have and continue to have access to an adequate number of subjects and the investigational device to complete the study.

The responsible monitor will write a report after each visit to the medical institutions. The reports will be sent to the sponsor and the principal clinical investigators.

Documentation and data processing Medical record of subjects

The following information should be clearly documented in medical record of subjects:

* That the subject is informed about the study and that the subject has signed the informed consent forms.
* That the subject is participating in the study; the identification code for the subject, the name of the study, and the study number (i.e., CREX-005).
* Which treatment the study refers to (i.e., C-REX Ring-locking Procedure with use of C-REX LapAid and C-REX DMH/DMHC).
* Name of the principal clinical investigator.
* All AEs and device deficiencies. Document and data control Prior to commencement of the study, clinical investigators and their staff will be informed about CIP, CRFs and other study documents and procedures.

For each subject enrolled, regardless of medical device initiation, a CRF must be completed and signed by corresponding investigation personnel. This applies to those subjects who fail to complete the study. If a subject withdraws from the study, the reason must be noted on CRF.

Data and information of subjects derived from the study are considered as source data. To ensure that all data are complete and correct, source data verification (SDV) will be confirmed by the monitor.

Comments in CRF should be made with a ballpoint pen with permanent ink in paper based CRF. In both paper based CRF and eCRF, if comments are missing in CRF, reasons for this must be stated. No questions, squares, fields or similar should be left without comments.

CRF entries and corrections will only be performed by investigational personnel, authorized by the principle clinical investigator. In paper based CRF, errors should be crossed out but not obliterated, the correction inserted, and the change initialled and dated by the clinical investigator.

Then entries will be checked by the monitor and any errors or inconsistencies will be checked and corrected immediately.

The responsible clinical investigator is obliged to keep the subject identification lists with the subject's identification code and identity in a safe place at the investigation site (hospital), accessible only to the investigation personnel. These source data and subject identification lists will be saved for 10 years after the close of the study at the medical institution.

NUMBER OF SUBJECTS The aim of this study is to verify the novel device in clinical practise in a big population. Since no control group is included, there is no need for power determinations.

Considering that similar anastomotic devices have been used in clinic for decades, the study will include about 250 subjects from 5 different centres/hospitals. In which, 100 subjects will be included in Fudan University Shanghai Cancer Center.

STATISTICAL ANALYSIS OF VARIABLES Descriptive methods are used to analyze the data collected in the study. The incidences of anastomotic leakage and other AEs/device deficiencies are calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥18 years and ≤80 years.
2. Planned resection due to benign or malign disease in the left colon (descending colon and sigmoid) or the upper rectum (15 cm above the anal rim).
3. Cognitive ability to take part in the study and understand the information he/she receives about participating in the study.
4. The patient has signed a written informed consent.

Exclusion Criteria:

1. Urgent medical condition requiring immediate care.
2. Current surgical conditions, such as intestinal obstruction or perforation, local or systemic infections, peritonitis, intestinal ischemia or severe dissemination (metastases) of cancer.
3. Stenosis or other obstructions in the anal passage.
4. Previous major abdominal surgery, previous radiation therapy to organs in abdomen or pelvis.
5. Health condition classified as ASA III - VI .
6. Albumin level less than 35 g/l.
7. Inflammatory bowel disease (IBD) (ulcerative colitis or Crohn´s disease).
8. Disease that requires more than one anastomosis during the surgical procedure.
9. Treatment with cortisone and/or other immunosuppressive medications less than one month before surgery.
10. Contraindications to general anaesthesia.
11. Perioperative detection of extreme variants of intestinal diameters or wall thickness.
12. Cognitive ability that limits the patient's ability to take part in the study and understand the information he/she received about participating in the study, or the patient does not agree to join the study.
13. BMI > 35.
14. Myocardial infarct ≤ 6 months or sever heart disease.
15. Severe embolic disease.
16. Other conditions which surgeons think the patient should be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence rate of complication related to the investigational device | Up to 30 days after surgery
  Complications related to the investigational device, for instance anastomotic leakage, anastomotic bleeding, excess fluid in abdominal drainage, CT scan verified abdominal abscess

SECONDARY OUTCOMES:
Time to evacuation of the short-term implant | About 2 weeks after surgery
  The subject informs the clinical investigator and hand over the expelled short-term implant
Time to first defecation | Up to 30 days after surgery
  The subject informs the clinical investigator when this occurs
Time to first intestinal sounds | Up to 30 days after surgery
  The subject informs the clinical investigator about when the intestine begin to murmur, and the clinical investigator will check the sound with a stethoscope
Time to passage of gas | Up to 30 days after surgery
  The subject informs the clinical investigator when it occurs
Number of postoperative interventions related to the investigational device | Up to 30 days after surgery
  The clinical investigator notes the interventions after surgery related to the use of device, for instance, CT scan, endoscopy examination and re-operation etc
Anastomotic integrity pressure | The operation day
  To confirm that the two anastomotic rings are properly locked to each other, measure integrity pressure through catheters connected to DMC (if DMC is applied). By infusing air into the closed space adjacent to the anastomosis via on catheter and concomitantly camping the other three catheters. When the pressure in the closed space exceeds the contact-induced closure by the joined intestinal segments, the pressure abruptly dropped and is defined as integrity pressure
Time of surgery | The operation day
  The time to complete the operation

OTHER OUTCOMES:
Hemoglobin | Up to 30 days after surgery, when needed
  Blood tests to detect potential anastomotic leakage
WBC (white blood cell) | Up to 30 days after surgery, when needed
  Blood tests to detect potential anastomotic leakage
Physical examination | Up to 30 days after surgery
  Body temperature, palpation of abdomen etc
Procedures and/or device related adverse events | Up to 30 days after surgery
  The clinical investigator notes the adverse events, severity and the relation to the investigational device

CONTACTS AND LOCATIONS:
Overall Officials: Sanjun Cai, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No